CLINICAL TRIAL: NCT01262066
Title: RCT of LifeSkills Workshop on BP in Hypertensive Employees
Brief Title: Effects of Lifeskills Workshop on BP in Hypertensive Employees
Acronym: Lifeskills BP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Lynn Clemow, Ph.D., Williams LifeSkills, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lifeskills BP study; R44HL067584 (NIH)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2010-11

CONDITIONS: Hypertension
Keywords: hypertension; stress reduction
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LifeSkills workshop intervention (Experimental): Participants attended 10 1-hr weekly sessions. The content of the groups followed the LifeSkills Workshop manual and Video(Williams LifeSkills, Inc, Durham NC). The LifeSkills Workshop is a structured psycho-educational group intervention using workbooks and videotapes that draw on cognitive-behavioral techniques and stress reduction approaches.
  Interventions: Behavioral: Lifeskills Workshop Intervention
- Enhanced usual care (No Intervention): The Usual Care group received a self-help brochure on BP control developed by the National Heart, Lung, and Blood Institute (NHLBI). In addition, with the participants' permission, their BP readings were sent to their listed physicians, along with the 1-page JNC-7 express summary for the management of high BP.

INTERVENTIONS:
Behavioral: Lifeskills Workshop Intervention — Intervention participants attended 10 one-hour weekly group sessions. The content of the groups followed the LifeSkills Workshop manual and Video ( (Williams LifeSkills, Inc, Durham NC). The LifeSkills Workshop is a structured psycho-educational group intervention using workbooks and videotapes that draw on cognitive-behavioral techniques and stress reduction approaches.
  Arms: LifeSkills workshop intervention

SUMMARY:
A number of psychosocial risk factors have been strongly related to a range of health problems (chief among them CVD). Clinical research has shown that behavioral interventions have enormous promise to ameliorate the psychosocial distress, the health-damaging effects and the costs associated with these risk factors. However, few such programs have been implemented in a large-scale way. Corporations are increasingly interested in providing such services for their employees, but they have encountered difficulties in knowing which programs are most effective. Until these programs are developed as products that can be tested and shown to produce consistent benefits, dissemination of these beneficial programs will be hindered. Taken together, these findings make a strong case that the development of a standardized, protocol-driven behavioral intervention package that can be delivered in a wide range of corporate settings presents a remarkable commercial opportunity. The overall goal of this SBIR Fast-Track-funded project is to gain empirical evidence in a RCT that documents the effectiveness of the Williams LifeSkills Workshop (a protocol driven 6-session workshop) in reducing BP, psychosocial risk factors, and promoting positive health outcomes in a cost effective manner in a corporate setting. This empirical support, tested in a setting independent of the program developers and by an experienced research team, will then be used to help market the product in the corporate wellness marketplace. It is hypothesized that participants (employees in an urban medical center) in the LifeSkills intervention will experience greater reductions in blood pressure and improvements in measures of psychosocial well-being than those receiving usual medical care and given educational materials on reducing BP.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-75
* Employees of Columbia University Medical Center
* BP >= 140/90 on 2 occasions (average of 3 readings each time)

Exclusion Criteria:

* Pregnancy
* End-stage Renal disease
* BP > 165/110 (average over 3 readings)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2002-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
change in mean office BP, covarying hostility and hostility x time (stratification variable) | 2 months after end of treatment
  The change in the mean office BP (evaluated automatically by BP-Tru device) from baseline to follow-up. Hostility, evaluated by Cook-Medley questionnaire (Barefoot scoring) was a stratification variable and thus was used as a covariate in the analysis

SECONDARY OUTCOMES:
Changes in mean office BP, controlling for baseline medications and medication changes during trial | baseline to follow-up 2 months after end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lynn P Clemow, PhD, Principal Investigator — Columbia University